CLINICAL TRIAL: NCT06584032
Title: A Randomized,Open-label,Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of Fruquintinib Plus Sintilimab Versus Chemotherapy of the Treating Physician's Choice as Second-line Treatment for Advanced Endometrial Cancer
Brief Title: Study of Fruquintinib Plus Sintilimab for Treatment of Advanced Endometrial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-013-00CH1
Record Dates: First submitted 2024-08-21; First posted 2024-09-04 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Advanced Endometrial Cancer
Keywords: fruquintinib; sintilimab; endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — HMPL-013; sintilimab; Paclitaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will be treated with a planned dose of fruquintinib and sintilimab every three weeks until an IRC (independent review committee)-confirmed PD(disease progression) or meeting other discontinuation criteria.
  Interventions: Drug: fruquintinib; Biological: sintilimab
- Control group (Active Comparator): Patients will be treated with TPC (chemotherapy of treating physician's choice, paclitaxel or doxorubicin) every three or four weeks until IRC-confirmed PD or meeting other discontinuation criteria.
  Interventions: Drug: paclitaxel; Drug: doxorubicin

INTERVENTIONS:
Drug: fruquintinib — Fruquintinib will be orally administrated once daily for 2 consecutive weeks followed by a 1-week break.
  Other Names: HMPL-013
  Arms: Experimental group
Biological: sintilimab — Sintilimab will be intravenously administrated on Day 1 every three weeks.
  Other Names: IBI308
  Arms: Experimental group
Drug: paclitaxel — 175 mg/m^2 via IV infusion, once a week for 3 weeks followed by a 1-week break.
  Arms: Control group
Drug: doxorubicin — 60mg/m^2 via IV infusion, on Day 1 every three weeks.
  Arms: Control group

SUMMARY:
The goal of this study is to evaluate whether fruquintinib(HMPL-013) plus sintilimab(IBI308) is safe and effective in the treatment of advanced endometrial cancer(EMC).

DETAILED DESCRIPTION:
A randomized, open, positive-controlled, multicenter Phase III clinical study to compare the efficacy and safety of fruquintinib(HMPL-013) plus sintilimab(IBI308) versus chemotherapy in patients with advanced endometrial cancer who have progressed after first-line standard chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood and voluntarily signed the informed consent form
2. Age 18 to 75 years (inclusive) ; Body mass index (BMI) ≥ 18.5kg/m^2;
3. Histologically or cytologically confirmed advanced or recurrent endometrial cancer with measurable lesions
4. Patients who previously failed first-line systemic platinum-based therapy
5. ECOG PS (Eastern Cooperative Oncology Group performance status score) 0 or 1;
6. Need to provide tumor samples for central lab testing of biomarkers such as MSI(microsatellite instability) status;
7. Non-MSI-H(non-microsatellite instability-high) by central lab or previous test result indicating pMMR(proficient mismatch repair);
8. Adequate function of the major organs;
9. Expected survival ≥ 12 weeks;
10. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before randomization.

Exclusion Criteria:

1. Endometrial carcinosarcoma or sarcoma;
2. Known MMR(mismatch repair)/MSI status with dMMR(deficient mismatch repair) or MSI-H(microsatellite instability-high);
3. Toxicities related to prior anticancer therapy did not recover to ≤CTCAE Grade 1, except alopecia and oxaliplatin-induced peripheral neurotoxicity ≤CTCAE Grade 2;
4. Received systemic anti-tumor therapy approved within 4 weeks before randomization;
5. Other malignancies within the past 5 years;
6. Previous or screening central nervous system (CNS) metastases;
7. Radical radiotherapy within 4 weeks before randomization
8. Previously received any anti-programmed cell death receptor-1 (PD-1) antibody, anti-PD-L1(programmed death ligand-1) antibody, anti-PD-L2(programmed death ligand-2) antibody, or anti cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibody or any other antibody acting on T cell costimulation or checkpoint pathways (eg, OX40, CD137, etc) or small molecule vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitors;
9. Symptomatic or treatment-requiring thyroid dysfunction at screening;
10. Use of immunosuppressive agents within 4 weeks before randomization
11. Presence of any active autoimmune disease requiring systemic treatment or history of autoimmune disease within the past 2 years;
12. Systemic immunostimulants within 4 weeks before randomization;
13. Administration of any live or live-attenuated vaccine within 4 weeks before randomization or planned during the study;
14. Major surgical procedures within 4 weeks before randomization;
15. Uncontrolled malignant pleural effusion, ascites or pericardial effusion;
16. Patients with current hypertension uncontrolled by medication;
17. Patients with any current disease or condition affecting drug absorption, or patients unable to take oral medications;
18. Receiving strong inducers of cytochrome P450 3A4 enzyme;
19. Patients with gastrointestinal diseases or unresected tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding and perforation as judged by the investigator; or with gastrointestinal perforation or gastrointestinal fistula, which is not recovered after surgical treatment;
20. Active bleeding within 3 weeks before randomization, or melena, or bleeding from a tumor within 2 weeks before the first dose ;
21. Tumor invading major vascular structures and is judged by the investigator to be at greater risk of massive haemorrhage;
22. Patients who had arterial thrombosis or deep venous thrombosis within 6 months before randomization; or patients who had stroke events and/or transient ischemic attack within 12 months; patients who had thrombosis caused by implantable intravenous infusion pump or catheter, except patients who had stable thrombosis after conventional anticoagulant therapy;
23. Clinically significant cardiovascular disease;
24. Clinically significant electrolyte abnormalities as judged by the investigator;
25. Active infection or fever of unknown origin before randomization;
26. Patients with active pulmonary tuberculosis (TB) receiving anti-tuberculosis treatment or anti-tuberculosis treatment within 1 year before randomization;
27. Patients with previous and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired pulmonary function, which may interfere with the detection and management of suspected drug-related pulmonary toxicity; previous or current (non-infectious) pulmonary inflammation requiring steroid hormone therapy;
28. Positive human immunodeficiency virus (HIV) antibody screening;
29. Known history of clinically significant liver disease
30. Known hypersensitivity to any of the study drugs or any of their excipients, or previous history of serious hypersensitivity to any other monoclonal antibody;
31. Patients who have received other clinical drugs that have not been approved or marketed within 4 weeks before randomization;
32. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
33. Patients who have received tissue/organ transplantation;
34. Patients with known psychiatric disorders or substance abuse disorders that could affect study compliance;
35. Patients who, in the opinion of the investigator, have other reasons that would make them inappropriate for this clinical study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-01-08 (Estimated); Study Completion 2029-06-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as assessed by IRC | Up to approximately 4 years
  Progression-free survival (PFS) is defined as the time from randomization to disease progression assessed by IRC or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 4 years
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 4 years
  Objective Response Rate (ORR) is defined as the ratio of patients who reached complete response (CR) or partial response (PR) , as assessed by IRC and investigator.
Duration of Response (DoR) | Up to approximately 4 years
  For patients who reached complete response (CR) or partial response (PR), Duration of Response (DoR) is defined as the time from the first CR or PR until disease progression or death due to any cause, whichever occurs first ,as assessed by IRC and investigator.
Disease Control Rate (DCR) | Up to approximately 4 years
  Disease Control Rate (DCR) is defined as the ratio of patients who reached complete response (CR) or partial response (PR) or maintained a stable disease, as assessed by IRC and investigator.
Time To Response (TTR) | Up to approximately 4 years
  Time To Response (TTR) is defined as the time from the start of treatment to the first objective response rate (ORR) ,as assessed by IRC and investigator.
Progression-Free Survival (PFS) as assessed by investigator | Up to approximately 4 years
  Progression-Free Survival is defined as the time from randomization to disease progression assessed by investigator or death due to any cause, whichever occurs first.
Incidence and severity of Treatment-emergent Adverse Events (TEAE) | Up to approximately 4 years
  Adverse events classified according to NCI CTCAE version 5.0
Blood concentration of fruquintinib | At the end of cycle 4 day 14 (each cycle is 21 days)
  Steady-state blood concentration of fruquintinib
Health-related quality of life (using EORTC QLQ-C30) | Up to approximately 4 years
  Changes in EORTC QLQ-C30(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) scores from baseline
Health-related quality of life (using EORTC QLQ-EN24) | Up to approximately 4 years
  Changes in EORTC QLQ-EN24 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Endometrial Cancer Module) scores from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Principal Investigator — Fudan University
Locations (17):
- China (17):
  - Beijing Obstetrics and Gynecology Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - SUN Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xijing Hospital of Air Force Military Medical University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sencond Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Women's Hospital school of Medical Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang